CLINICAL TRIAL: NCT03047746
Title: Unrelated And Partially Matched Related Donor Peripheral Blood Stem Cell Transplantation (PSCT) With TCR αβ + T Cell And B Cell Depletion For Patients With Acquired And Inherited Bone Marrow Failure
Brief Title: Unrelated And Partially Matched Related Donor PSCT w/ T Cell Receptor (TCR) αβ Depletion for Patients With BMF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Timothy Olson, Timothy Olson M.D. Ph.D., Assistant Professor Pediatrics, Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-012881
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Acquired Aplastic Anemia; Paroxysmal Nocturnal Hemoglobinuria; Inherited Bone Marrow Failure Syndromes
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Congenital Bone Marrow Failure Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- TCRalpha/beta Tcell Depletion for BMF with trilineage aplasia (Other): Patients with acquired or inherited bone marrow failure (iBMF) with trilineage aplasia excluding Fanconi Anemia will be given previously established, disease-specific chemotherapy and/or radiation based conditioning regimens prior to hematopoietic stem cell transplantation using TCRalpha/beta and B cell depleted peripheral blood stem cells from unrelated or partially matched related donors.
  Interventions: Device: CliniMACs
- TCRalpha/beta Tcell Depletion for BMF w/o trilineage aplasia (Other): Patients with acquired or inherited bone marrow failure (iBMF) without trilineage aplasia will be given previously established, disease-specific chemotherapy and/or radiation based conditioning regimens prior to hematopoietic stem cell transplantation using TCRalpha/beta and B cell depleted peripheral blood stem cells from unrelated or partially matched related donors.
  Interventions: Device: CliniMACs
- TCRalpha/beta Tcell Depletion for BMF w/ Fanconi Anemia (Other): Patients with acquired or inherited bone marrow failure (iBMF) with Fanconi Anemia and related DNA Repair Disorders will be given previously established, disease-specific chemotherapy and/or radiation based conditioning regimens prior to hematopoietic stem cell transplantation using TCRalpha/beta and B cell depleted peripheral blood stem cells from unrelated or partially matched related donors.
  Interventions: Device: CliniMACs

INTERVENTIONS:
Device: CliniMACs — Peripheral blood stem cells from closely matched unrelated or partially matched related donors will be processed using the CliniMACS device to remove TCRalpha/beta T cells and B cells, in accordance with the Investigator Brochure and Technical Manual following the laboratory standard operating procedures (SOPs) and using aseptic technique

SUMMARY:
This is a single arm pilot study using TCR alpha/beta+ T cell-depleted peripheral blood stem cells (PBSC) from closely matched unrelated donors or partially matched/haploidentical related donors for hematopoietic stem cell transplant (HSCT) in patients with acquired and inherited bone marrow failure (BMF) syndromes.

DETAILED DESCRIPTION:
This is a single arm pilot study using TCR alpha/beta+ T cell-depleted peripheral blood stem cells (PBSC) from closely matched unrelated donors or partially matched/haploidentical related donors for hematopoietic stem cell transplant (HSCT) in patients with acquired and inherited bone marrow failure (BMF) syndromes. Previously established, disease-specific transplant preparative regimens will be administered based on the specific underlying BMF condition. Mobilized PBSC will be processed using the CliniMACS system for TCR alpha/beta+ T cell depletion plus cluster of differentiation 19+ (CD19+) B cell depletion. The study will determine efficacy of this strategy in terms of engraftment, rates of acute and chronic Graft versus Host Disease (GvHD), and one year overall and event-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Acquired and Inherited Bone Marrow Failure Conditions Associated with Trilinear Bone Marrow Failure

  * Acquired Aplastic Anemia

    1. Must meet criteria for severe or very severe aplastic anemia (AA), defined by:

       i. Bone marrow biopsy demonstrating cellularity of <25% overall or bone marrow biopsy that is overall hypocellular for age by pathology report with reductions in any two hematopoietic lineages (myeloid, erythroid, or megakaryocyte)

       ii. In addition, 2 of the following must be met:
       1. absolute neutrophil count (ANC) < 500/µL (severe) or < 200/µL (very severe). Current ANC or last ANC prior to start of Granulocyte-colony stimulating factor (G-CSF) may be used.
       2. platelets < 30,000/µL or transfusion dependence
       3. absolute reticulocyte count < 40,000/µL

       iii. Negative evaluation for inherited bone marrow failure conditions (see below)

       iv. Must not have accompanying diagnosis of myelodysplastic syndrome
    2. Patients meeting other eligibility criteria may receive study therapy as the initial treatment approach provided an eligible unrelated or mismatched related ("haplo") donor is available
    3. Patients who have received prior immune suppression therapy will be eligible if they have refractory or relapsed disease defined as per treating clinician's judgement, at least 12 weeks after initiation of immune suppression therapy. Relapsed patients who previously met hematologic criteria for severe aplastic anemia do not have to meet these hematologic criteria for severe aplastic anemia at time of relapse to be eligible for transplant.
  * Paroxysmal Nocturnal Hemoglobinuria

    1. Patients must have testing (eg. Flow Cytometry demonstrating cells with absent cluster of differentiation 55 (CD55) or cluster of differentiation 59 (CD59) expression demonstrating a PNH clone in greater than 10% of peripheral blood red blood cells and/or granulocytes, along with clinical or laboratory evidence of intravascular hemolysis, such as:

       i. Elevated Lactate dehydrogenase (LDH)

       ii. Low to absent serum haptoglobin

       iii. Hemoglobinuria

       iv. Reticulocytosis

       v. Studies demonstrating aberrant complement activation
    2. Patients who have small paroxysmal nocturnal hemoglobinuria (PNH) clones, no evidence of hemolysis, and meet criteria for severe or very severe AA as defined above, will be classified as acquired AA for treatment stratification.
  * Fanconi Anemia

    1. To be eligible, patients must meet the following criteria:

       i. Must have evidence of BM failure, defined as a bone marrow biopsy demonstrating cellularity of <25% in addition to peripheral blood cytopenias

       ii. Must have chromosomal breakage (stress) testing performed demonstrating increased sensitivity to DNA damage caused by mitomycin C (MMC) or diepoxybutane (DEB)

       iii. Specific testing to define the subtype of Fanconi Anemia through genetic sequencing for causative mutations or complementation group studies is strongly recommended, though not required.
  * Dyskeratosis Congenita and related telomere disorders

    1. To be eligible, patients must meet the following criteria:

       i. Must have evidence of BM failure, defined as a bone marrow biopsy demonstrating cellularity of <25% in addition to peripheral blood cytopenias

       ii. Must have lymphocyte telomere length analysis performed at a Clinical Laboratory Improvement Amendments (CLIA)-certified facility, demonstrating telomeres <1%ile for age

       iii. Specific gene sequencing testing to define the causative genetic mutation is strongly recommended, though not required.
  * Shwachman-Diamond Syndrome

    1. To be eligible, patients must meet the following criteria:

       i. Must have genetic testing confirming a mutation in the Shwachman-Bodian-Diamond syndrome (SBDS) gene, and/or classic clinical features of Shwachman-Diamond Syndrome, including pancreatic insufficiency, musculoskeletal anomalies, and endocrinopathies

       ii. Must have developed trilineage BM failure, including BM cellularity < 25%.
    2. Patients meeting the above criteria for Shwachman-Diamond syndrome will be eligible for conditioning regimen #1 with dosing of Total Body Irradiation (TBI) and cyclophosphamide according to the dyskeratosis congenita regimen
* Inherited Bone Marrow Failure Conditions Associated with Predominant Single Lineage Failure

  * Severe Congenital Neutropenia

    1. To be eligible, patients must meet the following criteria:

    i. Have a baseline ANC < 500/µL prior to G-CSF therapy

ii. Require chronic G-CSF therapy greater than 3 doses per week in order to maintain an ANC > 1000/µL

iii. Have genetic testing demonstrating mutation(s) in a gene known to cause severe congenital neutropenia and/or have negative testing for autoimmune causes of neutropenia or BM biopsy demonstrating myeloid lineage arrest at neutrophil precursor stage.

iv. History of severe bacterial or fungal infection associated with neutropenia, including, but not limited to, pneumonia, osteomyelitis, mastoiditis, or bacteremia. If no infection history, must otherwise have evidence of toxicity due to chronic G-CSF therapy, including osteopenia, splenomegaly or isolated cytogenetic abnormalities.

* Isolated disorders of erythropoiesis:

  1. Includes, but not limited to: i. Diamond-Blackfan Anemia (DBA) ii. Congenital Dyserythropoietic Anemia (CDA) iii. Congenital Sideroblastic Anemia (CSA) 2. Eligibility criteria include: i. Chronic red blood cell (RBC) Transfusion Dependence, with minimum frequency of every 8 weeks ii. BM aspirate and biopsy demonstrating selective erythroid hypoplasia or dyserythropoiesis iii. For patients with DBA, must have failed at least one therapeutic trial with corticosteroids iv. Acquired viral and autoimmune causes of hypo-productive anemia have been excluded v. Specific genetic testing attempting to define the causative mutation is recommended but not required

  o Congenital Thrombocytopenia Syndromes

  1. Includes, but is not limited to, patients with Congenital Amegakaryocytic Thrombocytopenia caused by mutations in the MPL gene 2. Eligibility criteria include: i. Platelet transfusion dependence with a minimum transfusion frequency of every 8 weeks ii. Infectious, autoimmune, and other causes of secondary thrombocytopenia have been excluded iii. Genetic sequencing of the MPL gene is required iv. Additional genetic testing for causes of familial thrombocytopenia is recommended but not required
* Organ function status

  * Renal: Serum creatinine <1.5x upper limit of normal for age
  * Hepatic: Transaminases <500 upper limit of normal. Bilirubin <2.5 mg/dL, (unless elevation due to Gilberts disease or known hemolytic anemia).
  * Cardiac: shortening fraction >= 27%
  * Pulmonary: Diffusing Capacity (DLCO) >= 50% predicted in patients old enough to comply with pulmonary function testing (PFTs) or no baseline oxygen requirement for younger patients.
  * Lansky or Karnofsky performance >= 60
* Infectious disease criteria

  * No active, untreated infections
  * Patients with likely bacterial infections must be receiving appropriate antibacterial therapy and demonstrating therapy response
  * Patients with likely fungal infections must have had at least 2 weeks of appropriate anti-fungal antibiotics and be asymptomatic.
  * Patients with symptoms consistent with active viral infection will be deferred until viral symptoms resolve. Patients with evidence of cytomegalovirus (CMV), Epstein-Barr virus (EBV) or other known viremia must receive appropriate therapy to clear viremia prior to initiating study therapy.
* Signed consent by parent/guardian or able to give consent if >= 18 years

Exclusion Criteria:

* Patients who do not meet disease, organ or infectious criteria.
* Patients with a clinical diagnosis of myelodysplastic syndrome (MDS) defined by combination of bone marrow dysplasia and classic cytogenetic lesion (Monosomy 7, Trisomy 8 eg.), with or without excess blasts.
* Patients with no suitable closely Human leukocyte antigen (HLA)-matched unrelated or related haploidentical matched donor available. Patients with suitable fully matched related donor are also not eligible.
* Pregnant females. All females of childbearing potential must have negative pregnancy test.

Donor selection and eligibility:

• Donor selection will comply with 21 Code of Federal Regulations (CFR 1271) of the U.S. Food and Drug Administration's Code of Federal Regulations

Donor testing:

* Unrelated donor meets National Marrow Donor Program criteria for donation
* For partially matched related donors, Children's Hospital of Philadelphia (CHOP) bone marrow transplant (BMT) standard procedures apply for determining donor eligibility, including donor screening and testing for relevant communicable disease agents and diseases. The donor collection program is FACT accredited.
* For partially matched related donors, if subject has genetically confirmed iBMF syndrome, related donor must be evaluated for this disorder and testing must be negative
* Infectious disease testing of donor will be per current Blood and Marrow Transplant Program Standards of Practice as per 21 CFR Part 1271. Donor medical records and history are reviewed to confirm that the donor is free of infectious risk factors and meets donor eligibility criteria as defined by 21 CFR 127.

Donor matching

* High resolution HLA typing at HLA-A, -B, -C, DRB1, and DQB1 loci
* Unrelated donor
* Donor must be an antigen and allele match at ≥ 8/10 HLA Loci
* In donor with 2 mismatches, only one mismatch involving HLA-A, -B, or -DRB1 will be allowed
* Donor and collection center willing to undergo mobilization and apheresis
* Partially matched related donor
* Related donor must be ≥ 5/10 but < 10/10 HLA match
* Donor must be willing to undergo G-CSF mobilization and stem cell apheresis.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Rate of graft failure | Up to three years post-transplantation
Time to neutrophil engraftment | Up to 60 days post-transplantation
Incidence of acute graft vs. host disease (GVHD) | Up to 100 days post-transplantation
Incidence of chronic graft vs. host disease (GVHD) | Up to three years post-transplantation

SECONDARY OUTCOMES:
Treatment-related Mortality (TRM) | Up to 100 days post-transplantation
Probability of event-free survival (EFS) | Up to 1 year post-transplantation
Probability of overall survival (OS) | Up to 1 year post-transplantation
Reactivation/Infection from CMV, EBV, adenovirus | Up to 1 year post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Olson, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No